CLINICAL TRIAL: NCT01726946
Title: A Phase 2, Multicenter, Dose-Ranging Study to Evaluate the Safety and Efficacy of VX-135 With Ribavirin in Treatment-Naïve Subjects With Chronic Hepatitis C
Brief Title: A Phase 2 Study to Evaluate the Safety and Efficacy of VX-135 With Ribavirin in Treatment-Naïve Subjects With Chronic Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VX12-135-101
Record Dates: First submitted 2012-11-07; First posted 2012-11-15 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis C; HCV; CHC
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- VX-135 High Dose with ribavirin (Experimental): 12 weeks of a high dose of VX-135 in combination with ribavirin
  Interventions: Drug: VX-135; Drug: ribavirin
- VX-135 Low Dose with ribavirin (Experimental): 12 weeks of a low dose of VX-135 in combination with ribavirin
  Interventions: Drug: VX-135; Drug: ribavirin

INTERVENTIONS:
Drug: VX-135 — 12 weeks of VX-135
Drug: ribavirin — 12 weeks of ribavirin

SUMMARY:
A Phase 2 study to evaluate the safety and efficacy of two different once daily doses VX-135 in combination with ribavirin in treatment-naïve subjects with chronic hepatitis C

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects (male and female) must be between the ages of 18 and 60 years at screening
* Subjects must have genotype 1 Chronic Hepatitis C
* Subjects must be treatment naïve
* Subjects must have laboratory values at screening within limits as specified by the protocol

Key Exclusion Criteria:

* Evidence of cirrhosis
* Female subjects who are pregnant or nursing or male subjects with a female partner of childbearing potential who is unwilling to adhere to the contraception requirements, is pregnant or nursing, or planning to become pregnant during the study
* Any other cause of significant liver disease in addition to hepatitis C
* Human immunodeficiency virus -1 or -2
* Diagnosis of or suspected hepatocellular carcinoma
* History of organ transplant, with the exception of corneal transplants and skin grafts

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability as assessed by adverse events, vital signs, 12-lead electrocardiograms, echocardiograms (Cohorts 1 and 2 only), and laboratory assessments | Up to 52 weeks

SECONDARY OUTCOMES:
The proportion of subjects who have an SVR at 4 weeks after the last planned dose of treatment (SVR4) | 16 weeks
The proportion of subjects who have an SVR at 12 weeks after the last planned dose of treatment (SVR12) | 24 weeks
The proportion of subjects who have an SVR at 24 weeks after the last planned dose of treatment (SVR24) | 36 weeks
The proportion of subjects who have virologic relapse | Up to 52 weeks
Viral kinetics, as determined at different time points by the proportion of subjects who achieve: -Undetectable HCV RNA -<LLOQ HCV RNA | Up to 64 weeks
The proportion of subjects who have virologic breakthrough | Up to 52 weeks
  as measured by on-treatment HCV RNA values
The proportion of subjects who achieve SVR12 by IL-28B genotype (CC versus non-CC) | up to 28 weeks
The amino acid sequence of the nonstructural (NS)5B protein in subjects who fail treatment | Up to 60 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Vertex Pharmaceuticals Incorporated
Locations (6):
- United States (6):
  - California, La Jolla, California
  - Florida, Orlando, Florida
  - Georgia, Marietta, Georgia
  - Tennessee, Germantown, Tennessee
  - Texas, Arlington, Texas
  - Texas, Houston, Texas